CLINICAL TRIAL: NCT04701541
Title: Is the Perioperative Change in Ultrasound-based Diaphragmatic Inspiratory Amplitude Predictive of Postoperative Atelectasis: A Prospective Observational Study in Obese Patients Undergoing Bariatric Surgery
Brief Title: Perioperative Diaphragmatic Ultrasound as Predictive Index of Atelectasis in Bariatric Surgery
Acronym: ECODIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Alessandri, Principal Investigator, Level I Medical Director, MD, PhD, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECODIABAS
Record Dates: First submitted 2020-05-11; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pulmonary Atelectasis; Morbid Obesity
Keywords: Atelectasis; Diaphragmatic Inspiratory Amplitude; Obesity
MeSH Terms: conditions — Pulmonary Atelectasis; Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese Patients undergoing Bariatric Surgery (Other): Obesity is a progressively growing morbid condition in the world, and given the direct relationship between body mass index (BMI) and costs, this has a major impact on economic and health policy. Obese patients undergoing bariatric surgery are at high risk for postoperative respiratory complications. In these patients, postoperative respiratory complications are related to various pathophysiological mechanisms that include: decreased lung volumes, respiratory muscle dysfunction and atelectasis. Demographic (age, gender, BMI) and clinical features of the population included: ASA, comorbidity and pre and postoperative respiratory function [PaO2/FiO2, haemogasanalysis (EGA)]. Ultrasound evaluation of DIA was performed.
  T0: preoperative within 24h before surgery: DIA, haemogasanalysis; T1: Post operation: 60 min after extubation: Aldrete Score, DIA, EGA; T2: Post operation: 240 min after extubation: Aldrete, EGA.
  Interventions: Device: Diaphragmatic Ultrasound

INTERVENTIONS:
Device: Diaphragmatic Ultrasound — Diaphragmatic ultrasound is non-invasive, portable, quick to perform, with a linear relationship between diaphragmatic movement and inspired volume. In eligible patients, a preoperative baseline ultrasound evaluation of the diaphragm and lungs is accomplished. Evaluation will be performed by a single operator, blinded to the arterial blood gas analysis values. In a semi recumbent position, patients will be asked to rest and breath quietly. An anterior approach will be carried out applying freehand transducer on abdomen at the right midclavicular line immediately below the costal margin with firm pressure, steering in cranial direction. A B-mode transverse scanning will be performed looking across the liver with gallbladder in the middle. Measurements will be recorded by the M-mode frozen images. The M-mode modality will be used to study DIA. The best sinusoidal curve will be considered for measurements.
  Other Names: Ultrasound-based Diaphragmatic Inspiratory Amplitude, ECO-DIA

SUMMARY:
In this study the Authors assume that peri-operative changes in DIA are predictive of postoperative atelectasis, thus providing a clinically useful tool to stratify the need for high-intensity monitoring, including admission to intensive care. Aim of this prospective observational study, in obese patients undergoing sleeve gastrectomy, is to evaluate the relationship between pre to postoperative changes in US-DIA and PaO2/FiO2.

DETAILED DESCRIPTION:
Obese patients undergoing bariatric surgery, are at high risk for postoperative respiratory complications but predictive variables, risk factors and criteria for postoperative ICU admission are debated. In these patients, postoperative respiratory complications are related to various pathophysiological mechanisms that include: decreased lung volumes, respiratory muscle dysfunction and atelectasis. Very recently it has also been demonstrated a possible role of molecules that would mediate the fibro-adipogenic remodeling of the diaphragm in the obese, thus increasing the respiratory disability.

Pulmonary atelectasis appears within minutes after anesthesia induction, complicate 85-90% of the cases -involving up to 15% of the lungs and inducing a 5 to 10% of cardiac output intra pulmonary shunting- and determine an increased incidence of postoperative morbidity (with higher incidence of pneumonia). Furthermore, in the perioperative period, obese patients are more likely to develop atelectasis that resolves more slowly than in non-obese patients. Surgical handling of sub diaphragmatic region, as during sleeve gastrectomy, can impair diaphragmatic excursions thus contributing to postoperative pulmonary dysfunction. The same upper abdominal surgery represents a risk factor for the development of pulmonary complications in the perioperative period and alteration of the respiratory function indices.

Ultrasounds (US) imaging is a real-time, bedside, non-invasive technique that allows the quantitative evaluation of amplitude, force and velocity of diaphragmatic movement, including: diaphragmatic inspiratory amplitude (DIA) and diaphragmatic thickening. The US-DIA is a qualified quantitative approach to assess diaphragmatic function and has been reported to linearly correlate with vital capacity. Recent studies have also correlated diaphragmatic dysfunction, which reduces the ability to generate total current volume, with the onset of atelectasis, but in a very specialized and dedicated area such as thoracic surgery. The originality of the study lies in the fact that the investigators have translated this method of evaluation of diaphragmatic function, as a predictive index of pulmonary complications in postoperative surgery, into a highly selected and clinically demanding type of patient, such as the patient suffering from pathological obesity.

Several guidelines have been created at European level for the perioperative management of the obese patient. One of the most recent is the one created by the Italian Society of Anaesthesia Analgesia Rianimazione e Terapia Intensiva (SIAARTI), which commissioned an "Obesity Task Force" of the Airway Management Study Group to coordinate a multidisciplinary multi-professional consensus project to identify bundles of Good Clinical Practices (GCPs), useful to define the risks in adult obese patients in hospital.

In obese patients undergoing sleeve gastrectomy there are no conclusive criteria for discharge and indications to postoperative ICU admission, as recently defined for patients with OSAS, the investigators hypothesize that perioperative change in US-DIA predicts postoperative atelectasis, thus providing a clinically useful tool to stratify the need for higher intensity monitoring including ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity undergoing bariatric surgery (BMI >30 Kg/m2)

Exclusion Criteria:

* Heart Failure
* Neuromuscular Diseases
* Previous Thoracic Surgery,
* American Society of Anesthesiology physical (ASA) status >III.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between diaphragmatic excursion and post-operative atelectasis | 240 minutes
  to detect the relationship between perioperative changes in DIA, (unit of measurement "millimeters") finally expressed as percentage differences at the baseline, during forced breath and occurrence and severity of postoperative atelectasis (evaluated through PaO2/FiO2 R) at 240 min after extubation (T2), view with haemogasanalytic measurement.

SECONDARY OUTCOMES:
amount of neuromuscular blockers | During surgery
  concentration of myorelaxants, expressed in milligrams, used during surgery. Measurement tool is the TOF Ratio [TOF Ratio, is the ratio of the amplitude of the fourth muscle response to the amplitude of the first]. Monitoring guide acceleromyographic train-of-four stimulus to the adductor pollicis.
difference in pre and postoperative DIA during calm breathing | During surgery + 1 hour post-surgery
  Quantification of the difference in diaphragmatic excursion, DIA (unit of measurement "millimeters") finally expressed as percentage differences at the baseline, during calm breathing between the pre-operative T0 time and the T1 time at 1 hour after the end of the operation.
incidence rate of pneumonia on the second postoperative day | 2 days
  The detection of pneumonia was carried out with CURB-65, a simple predictive clinical score based on mental confusion, azotemia (mg/dL), respiratory rate (n breaths/min), blood pressure (mmHg) and age (years). In addition, a chest X-ray was performed to highlight the presence of infiltrations.
hospitalization duration | 4 days
  average length of hospital stay in the post-operative period, in the general surgery department.
need for hospitalization in postoperative ICU | 4 days
  % of the patients need recovery in intensive care due to the onset of a complication during the post-operative course.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Alessandri, Principal Investigator — Emergency and Acceptance Depart., Anaesth. and Critical Areas, P. Umberto I
Locations (1):
- Hospital Policlinico Umberto I of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rose DK, Cohen MM, Wigglesworth DF, DeBoer DP. Critical respiratory events in the postanesthesia care unit. Patient, surgical, and anesthetic factors. Anesthesiology. 1994 Aug;81(2):410-8. doi: 10.1097/00000542-199408000-00020. PMID 8053592
- [Background] Chung F, Mezei G, Tong D. Pre-existing medical conditions as predictors of adverse events in day-case surgery. Br J Anaesth. 1999 Aug;83(2):262-70. doi: 10.1093/bja/83.2.262. PMID 10618941
- [Background] Members of the Working Party; Nightingale CE, Margarson MP, Shearer E, Redman JW, Lucas DN, Cousins JM, Fox WT, Kennedy NJ, Venn PJ, Skues M, Gabbott D, Misra U, Pandit JJ, Popat MT, Griffiths R; Association of Anaesthetists of Great Britain; Ireland Society for Obesity and Bariatric Anaesthesia. Peri-operative management of the obese surgical patient 2015: Association of Anaesthetists of Great Britain and Ireland Society for Obesity and Bariatric Anaesthesia. Anaesthesia. 2015 Jul;70(7):859-76. doi: 10.1111/anae.13101. Epub 2015 May 7. PMID 25950621
- [Background] Buras ED, Converso-Baran K, Davis CS, Akama T, Hikage F, Michele DE, Brooks SV, Chun TH. Fibro-Adipogenic Remodeling of the Diaphragm in Obesity-Associated Respiratory Dysfunction. Diabetes. 2019 Jan;68(1):45-56. doi: 10.2337/db18-0209. Epub 2018 Oct 25. PMID 30361289
- [Background] Duggan M, Kavanagh BP. Pulmonary atelectasis: a pathogenic perioperative entity. Anesthesiology. 2005 Apr;102(4):838-54. doi: 10.1097/00000542-200504000-00021. PMID 15791115
- [Background] Asteriou C, Lazopoulos A, Rallis T, Gogakos AS, Paliouras D, Barbetakis N. Fast-track rehabilitation following video-assisted pulmonary sublobar wedge resection: A prospective randomized study. J Minim Access Surg. 2016 Jul-Sep;12(3):209-13. doi: 10.4103/0972-9941.183483. PMID 27279390
- [Background] Reber A, Engberg G, Sporre B, Kviele L, Rothen HU, Wegenius G, Nylund U, Hedenstierna G. Volumetric analysis of aeration in the lungs during general anaesthesia. Br J Anaesth. 1996 Jun;76(6):760-6. doi: 10.1093/bja/76.6.760. PMID 8679345
- [Background] Brismar B, Hedenstierna G, Lundquist H, Strandberg A, Svensson L, Tokics L. Pulmonary densities during anesthesia with muscular relaxation--a proposal of atelectasis. Anesthesiology. 1985 Apr;62(4):422-8. doi: 10.1097/00000542-198504000-00009. PMID 3885791
- [Background] Gunnarsson L, Tokics L, Gustavsson H, Hedenstierna G. Influence of age on atelectasis formation and gas exchange impairment during general anaesthesia. Br J Anaesth. 1991 Apr;66(4):423-32. doi: 10.1093/bja/66.4.423. PMID 2025468
- [Background] Kelkar KV. Post-operative pulmonary complications after non-cardiothoracic surgery. Indian J Anaesth. 2015 Sep;59(9):599-605. doi: 10.4103/0019-5049.165857. PMID 26556919
- [Background] Eichenberger A, Proietti S, Wicky S, Frascarolo P, Suter M, Spahn DR, Magnusson L. Morbid obesity and postoperative pulmonary atelectasis: an underestimated problem. Anesth Analg. 2002 Dec;95(6):1788-92, table of contents. doi: 10.1097/00000539-200212000-00060. PMID 12456460
- [Background] Simonneau G, Vivien A, Sartene R, Kunstlinger F, Samii K, Noviant Y, Duroux P. Diaphragm dysfunction induced by upper abdominal surgery. Role of postoperative pain. Am Rev Respir Dis. 1983 Nov;128(5):899-903. doi: 10.1164/arrd.1983.128.5.899. PMID 6638679
- [Background] Dureuil B, Desmonts JM, Mankikian B, Prokocimer P. Effects of aminophylline on diaphragmatic dysfunction after upper abdominal surgery. Anesthesiology. 1985 Mar;62(3):242-6. doi: 10.1097/00000542-198503000-00006. PMID 3977111
- [Background] Manikian B, Cantineau JP, Bertrand M, Kieffer E, Sartene R, Viars P. Improvement of diaphragmatic function by a thoracic extradural block after upper abdominal surgery. Anesthesiology. 1988 Mar;68(3):379-86. doi: 10.1097/00000542-198803000-00010. PMID 3344992
- [Background] Nguyen NT, Lee SL, Goldman C, Fleming N, Arango A, McFall R, Wolfe BM. Comparison of pulmonary function and postoperative pain after laparoscopic versus open gastric bypass: a randomized trial. J Am Coll Surg. 2001 Apr;192(4):469-76; discussion 476-7. doi: 10.1016/s1072-7515(01)00822-5. PMID 11294404
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Kantarci F, Mihmanli I, Demirel MK, Harmanci K, Akman C, Aydogan F, Mihmanli A, Uysal O. Normal diaphragmatic motion and the effects of body composition: determination with M-mode sonography. J Ultrasound Med. 2004 Feb;23(2):255-60. doi: 10.7863/jum.2004.23.2.255. PMID 14992363
- [Background] Ayoub J, Cohendy R, Dauzat M, Targhetta R, De la Coussaye JE, Bourgeois JM, Ramonatxo M, Prefaut C, Pourcelot L. Non-invasive quantification of diaphragm kinetics using m-mode sonography. Can J Anaesth. 1997 Jul;44(7):739-44. doi: 10.1007/BF03013389. PMID 9232305
- [Background] Ayoub J, Cohendy R, Prioux J, Ahmaidi S, Bourgeois JM, Dauzat M, Ramonatxo M, Prefaut C. Diaphragm movement before and after cholecystectomy: a sonographic study. Anesth Analg. 2001 Mar;92(3):755-61. doi: 10.1097/00000539-200103000-00038. PMID 11226114
- [Background] Cohen E, Mier A, Heywood P, Murphy K, Boultbee J, Guz A. Excursion-volume relation of the right hemidiaphragm measured by ultrasonography and respiratory airflow measurements. Thorax. 1994 Sep;49(9):885-9. doi: 10.1136/thx.49.9.885. PMID 7940428
- [Background] Lloyd T, Tang YM, Benson MD, King S. Diaphragmatic paralysis: the use of M mode ultrasound for diagnosis in adults. Spinal Cord. 2006 Aug;44(8):505-8. doi: 10.1038/sj.sc.3101889. Epub 2005 Dec 6. PMID 16331304
- [Background] Blaivas M, Brannam L, Hawkins M, Lyon M, Sriram K. Bedside emergency ultrasonographic diagnosis of diaphragmatic rupture in blunt abdominal trauma. Am J Emerg Med. 2004 Nov;22(7):601-4. doi: 10.1016/j.ajem.2004.08.015. PMID 15666270
- [Background] Kim SH, Na S, Choi JS, Na SH, Shin S, Koh SO. An evaluation of diaphragmatic movement by M-mode sonography as a predictor of pulmonary dysfunction after upper abdominal surgery. Anesth Analg. 2010 May 1;110(5):1349-54. doi: 10.1213/ANE.0b013e3181d5e4d8. PMID 20418298
- [Background] American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Practice guidelines for the perioperative management of patients with obstructive sleep apnea: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Anesthesiology. 2014 Feb;120(2):268-86. doi: 10.1097/ALN.0000000000000053. No abstract available. PMID 24346178

DOCUMENTS (3):
  • Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT04701541/SAP_000.pdf
  • Study Protocol (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT04701541/Prot_001.pdf
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT04701541/ICF_002.pdf